CLINICAL TRIAL: NCT01708330
Title: The Effect of Topical Lidocaine on Pain Scores During Manual Vacuum Aspiration for Nonviable Pregnancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bridgeport Hospital (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Amanda Tower, Fellow, Bridgeport Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-0039
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Nonviable Pregnancy
Keywords: manual vacuum aspiration; missed abortion; incomplete abortion; nonviable pregnancy; topical lidocaine
MeSH Terms: conditions — Abortion, Missed; Abortion, Incomplete | interventions — Lidocaine; K-Y jelly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo gel (Placebo Comparator): Placebo gel applied topically to the cervix
  Interventions: Drug: Placebo gel
- Lidocaine gel (Experimental): 2% lidocaine gel applied topically to the cervix
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — 2% Lidocaine gel
  Arms: Lidocaine gel
Drug: Placebo gel — odorless, colorless gel will be used as a placebo
  Other Names: KY Jelly
  Arms: Placebo gel

SUMMARY:
When a patient requires a manual vacuum aspiration (MVA), whether for an undesired pregnancy, missed abortion, or other nonviable pregnancy, she is undergoing an emotional experience. She is grieving the loss of her pregnancy, and is then faced with the anxiety of an invasive and often painful procedure. Minimizing the pain during this procedure must not be overlooked. There have been no randomized controlled trials evaluating pain control during MVA for nonviable pregnancy, and the data is mixed regarding analgesia for MVA for an elective abortion or other office procedures.

Women being treated at the Women & Infants Triage who have experienced a first trimester missed abortion, inevitable abortion, incomplete abortion or other nonviable pregnancy and are being treated with an outpatient manual vacuum aspiration will be asked to enroll in this study. Those who wish to participate will be randomly assigned to treatment with lidocaine gel or a placebo gel applied to the cervix during their procedure.

The hypothesis is that topical lidocaine will decrease pain during manual vacuum aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Women and Infants Triage/Women's Emergency Department
* Vital signs are stable
* Ages 18 and older
* Have a missed abortion, inevitable abortion, incomplete abortion or other nonviable pregnancy
* Estimated gestational age up to 10 weeks
* Undergoing MVA at the Women and Infants Triage/Women's Emergency Department
* Able to read English or Spanish
* Able to give informed consent for involvement in the study

Exclusion Criteria:

* Allergic to lidocaine, iodine or betadine
* Known sensitivity to any component of the lidocaine or placebo gel.
* In acute distress
* Unable to give informed consent
* Unable to read English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pain during intracervical block | immediate
  Pain on visual analogue scale

SECONDARY OUTCOMES:
Pain during tenaculum placement | immediate
  Pain on visual analogue scale
Pain during cervical dilation | immediate
  Pain on visual analogue scale
Pain during uterine aspiration | immediate
  Pain on visual analogue scale

OTHER OUTCOMES:
Complications | 1 hour after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Infants Hospital Triage, Providence, Rhode Island, United States